CLINICAL TRIAL: NCT05213858
Title: Biological Markers for Post-Traumatic Stress Disorder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 178-21
Record Dates: First submitted 2022-01-16; First posted 2022-01-28 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Functional Neuroimaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CAPS questionnaire — PTSD diagnosis and severity will be done using the CAPS-5 questionnaire.
Diagnostic Test: Beck Depression Inventory — depression symptoms will be measured by the BDI-II. The BDI-II consists of 21 items and uses a 0 to 3 severity scale. Total scores range from 0 to 63, with higher scores indicating more severe depression.
Diagnostic Test: The Fibromyalgia Impact Questionnaire — The FIQ was developed from information gathered from patient reports, functional status instruments and clinical observations. This instrument measures physical functioning, work status (missed days of work and job difficulty), depression, anxiety, morning tiredness, pain, stiffness, fatigue and well-being over the past week.
Diagnostic Test: The Pittsburgh Sleep Quality Index — sleep patterns will be measured using the PSQI. This index assesses the quality and patterns of sleep in adults. It differentiates "poor" from "good" sleep quality by measuring seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, the use of sleeping medications and daytime dysfunction over the last month. Items are rated using a 0 to 3 scale. The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Diagnostic Test: Depression, Anxiety and Stress Scale-21 items — The DASS-21 is a three-scale self-report questionnaire designed to measure the emotional state of depression, anxiety and stress. Each scale contains 7 items, divided into subscales with similar content. Scores range between 0 and 21 in each subcategory.
Diagnostic Test: Traumatic Events Questionnaire — The TEQ examines experiences of traumatic events (e.g. sexual abuse, accidents and crime) that are considered potential triggers of PTSD symptoms. To assess trauma intensity, respondents provide information for each event that was experienced, as well as their age at the time of the event. The items are measured on a 9-point Likert scale from "not at all" to "severely/extremely". The TEQ has previously been used in Israel.
Diagnostic Test: Clinician Administered Dissociative States Scale — The CADSS is a 28-item structured clinical interview to assess state dissociation.
Diagnostic Test: A diary will be used for seven consecutive nights — A diary will be used for seven consecutive nights for the evaluation of:
  * Mean sleep latency
  * The number and duration of awakenings.
  * Subjective total sleep time
  * Subjective wake after sleep onset
  * Sleep efficiency
Diagnostic Test: MRI — Brain imaging will include DTI and resting state for structural and functional MRI scanning. Images will be acquired on MAGNETOM Vida 3T Scanner, configured with 64-channel receiver head coils (Siemens Healthcare, Erlangen, Germany) at the Department of Radiology at Shamir Medical Center.
Diagnostic Test: Functional brain imaging — Functional magnetic resonance imaging (fMRI) is widely used to study the operational organization of the human brain. This technology measures brain activity by detecting changes associated with blood oxygenation, using blood-oxygen-level-dependent imaging (BOLD) contrast.
Diagnostic Test: EEG analysis — EEG will be obtained using a point-of care device that consists of an EEG-Sense Headset, EEG-Sense Single-Use brush sensors, a pneumatic sensor positioning mechanism, EEG sampling electronics and software. The EEG-Sense Headset is an EEG electrode positioning system that quickly places electrodes in a uniform and consistent manner, to transfer electrophysiological EEG signals from an individual to a suitable EEG data collection device. The device is nonsterile, non-invasive and non-radiation emitting, and was developed for use in healthcare facilities and hospitals. Typical set-up and procedure time is several minutes. The device does not contain biologics, drugs, coatings or any claim of sterility. The EEG-Sense Single-Use brush sensors are made from well-established medical-grade materials; the Headset is made from Nylon 101. Electronic components and harnesses are embedded between two layers of nylon and are attached to each electrode port.
Diagnostic Test: Autonomic nervous system monitors — Data will be collected using Empatica's E4 wristband. Each of the study participants will wear the wristband for 7 days.
  Data collected from the band will include:
  ACC - Data from 3-axis accelerometer sensor in the range [-2g, 2g]. (sampled at 32 Hz) BVP - Data from photoplethysmography (PPG). (sampled at 64 Hz) EDA - Data from the electrodermal activity sensor in μS. (sampled at 4 Hz) IBI - Inter-beat intervals. (intermittent output with 1/64 second resolution) TEMP - Data from temperature sensors, expressed in degrees on the Celsius (°C) scale. (sampled at 4 Hz)

SUMMARY:
The current study aims to evaluate the sensitivity and specificity of a combination of various objective biomarkers for the diagnosis of PTSD.

DETAILED DESCRIPTION:
PTSD affects a major fraction of military combatants and is also very common in the general population. Like other psychiatric conditions, the diagnosis of PTSD is currently based on an interview and questionnaires. However, the validity of these tools is limited since it depends on the evaluator's skills, and on patient compliance and mental status; and may be prone to exaggeration or minimization of symptoms. This prompts an urgent need for evaluation that will combine biomarkers for objective diagnosis, and follow up of individuals with PTSD.

Knowledge has grown in recent years regarding the biologic pathophysiological cascade responsible for the development of a "non-healing wound in the brain" that characterizes PTSD. Shortly after the traumatic experience, fundamental changes in autonomic nervous and endocrine activity are evident, together with changes in brain function; these can become chronic in those with long-standing unremitting PTSD. Several studies indicate good correlations of the diagnosis and severity of PTSD, with objective biological measures such as heart rate variability (HRV), brain connectivity and endocrine activity. However, the currently available data on these biological variables are still not sufficient to be used for diagnosis of PTSD.

The aim of the current study is to characterize the biological fingerprint of PTSD, by using a combination of biological measures, for an objective diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. The willingness and ability to read, understand and sign an informed consent form.
2. Age 20-60 years.
3. A history of more than 2 years of combat service, and of at least one potentially life-threatening combat experience.
4. One year or more after the last combat experience.

Exclusion Criteria:

1. Inability to attend scheduled clinic visits or comply with the study protocol
2. A history of traumatic brain injury or any other known brain pathology.
3. Substance use, except for prescribed cannabis, if it can be withheld for at least 24 hours prior to the study evaluation.
4. A current psychiatric disorder other than PTSD.
5. The inability to perform an awake brain MRI.

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Male combatants aged 20-60 years, with a history of exposure to an apparently life threatening-combat event, with or without PTSD.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
correlation between CAPS score and mean heart rate variability | at baseline
  the correlation between CAPS score and mean heart rate variability will be evaluated

SECONDARY OUTCOMES:
correlation between CAPS score and fronto-limbic connectivity | at baseline
  the correlation between CAPS score and fronto-limbic connectivity will be evaluated using DTI
correlation between CAPS score and frontal activity | at baseline
  the correlation between CAPS score and frontal activity will be evaluated using BOLD MRI
correlation between CAPS score and depression score | at baseline
  the correlation between CAPS score and depression score will be evaluated using back depression inventory

CONTACTS AND LOCATIONS:
Overall Officials: keren doenyas-barak, md, Principal Investigator — sagol center for hyperbaric medicine
Locations (1):
- Assaf-Harofeh Medical Center, Ramla, Israel

IPD SHARING:
Plan to Share IPD: Undecided